CLINICAL TRIAL: NCT04591821
Title: Bowel Dysfunction 3 Years After Anterior Resection a in a Swedish National Cohort
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/992
Record Dates: First submitted 2020-09-15; First posted 2020-10-19 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Low Anterior Resection Syndrome; Rectal Cancer
MeSH Terms: conditions — Low Anterior Resection Syndrome; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objectives are to evaluate the prevalence of LARS and Quality of Life in rectal cancer patients 3 years after anterior resection, to investigate if anastomotic technique is a risk factor for major LARS and to study the prevalence of colostomy 3 years after anterior resection and evaluate stoma function according to the stoma scale in EORTC QLQ-CR29.

DETAILED DESCRIPTION:
All patients who have undergone anterior resection for rectal cancer between Q1 2015 and Q4 2017 have been identified in the Swedish Colorectal Cancer Registry (SCRCR). Three years after surgery the patients were sent a questionnaire including the LARS (Low Anterior Resection Syndrome)-score, the quality of life questionnaire EORTC QLQ 30 and CR29 in addition to a questionnaire regarding prevalence of remaining stoma.The patient cohort will be divided into two groups operated with total (TME) or partial (PME) mesorectal excision for further analyses. Patients with a stoma will be analysed separately.

Prevalence of major LARS and Quality of Life, QoL, 3 years after anterior resection will be assessed by the EORTC QLQ-C30 and by calculation of LARS Score with categories "no" (0-20 points), "minor" (21-29) and "major" (30-42). The LARS score will be dichotomized into the categories no/minor and major LARS.

Stoma function will be evaluated by the stoma scale in EORTC QLQ-CR29.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of rectal cancer in Sweden
* Operated on with anterior resection between Q1 2015 and Q4 2017 in Sweden, with or without defunctioning stoma

Exclusion Criteria:

* Age <18 years
* Dementia,
* Unable to understand Swedish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with rectal cancer that have undergone anterior resection for rectal cancer between Q1 2015 and Q4 2017 in Sweden
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Low Anterior Resection Syndrome score ( LARS Score) | 3 years
  Prevalence of low anterior resection syndrome (LARS) 3 years after low anterior resection for rectal cancer, assessed by the validated instrument LARS score consisting of 5 questions with a total score of between 4 and 42. .0-20 corresponds to no LARS, 21-29 to minor LARS and 30-42 to major LARS.
QoL | 3 years
  Quality of life measured by the validated EORTC (European Organisation for Research and Treatment of Cancer) questionnaires QLQ 30 (Quality of life questionnaire 30) consisting of 30 questions and CR 29 (colirecti 29), a specific questionnaire assessing quality of life in colorectal cancer patients, consisting of 29 questions. Both QLQ 30 and CR 29 include symptom scales and functional scales from 0-100 with lower scores on symptom scales indicating better quality of life and higher scores on functional scales indicating better quality of life.

SECONDARY OUTCOMES:
Correlation LARS score QoL | 3 years
  Correlation between low anterior resection syndrome (LARS) assessed by the validated instrument LARS score consisting of 5 questions with a total score of between 4 and 42, 0-20 corresponding to no LARS, 21-29 to minor LARS and 30-42 to major LARS, and the bowel dysfunction scale in EORTC (European Organisation for Research and Treatment of Cancer) questionnaire CR29 (colirecti 29) consisting of 6 questions with a total score between 6 and 24 with higher score indicating worse function.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Louise Lydrup, Assoc prof, Principal Investigator — Dept of surgery, Skåne university hospital, Malmö, Sweden
Locations (1):
- Skane university hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No